CLINICAL TRIAL: NCT00338026
Title: A Phase I, Dose Finding, Pharmacokinetic, and Safety Study of Continuous IV Infusion of ECO-4601 in Patients With Advanced Cancer Including an Extension Portion to Obtain Safety Data at the Highest Tolerable Dose
Brief Title: A Phase I Study of ECO-4601 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thallion Pharmaceuticals (Industry)
Responsible Party: Didier Reymond, MD / Vice-President Medical and Clinical Affairs, Thallion Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECO-4601-101
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Tumors; Glioma; Colorectal Cancer; Lung Cancer; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer
Keywords: Solid Tumors; Thallion; TLN-4601; Ecopia; ECO-4601; Patients with histologically confirmed solid tumors:; High Grade Glioma; Colorectal; Lung; Breast; Ovarian; Pancreatic; Prostate
MeSH Terms: conditions — Neoplasms; Glioma; Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — diazepinomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECO-4601 (Experimental)
  Interventions: Drug: ECO-4601

INTERVENTIONS:
Drug: ECO-4601 — Continuous IV infusion for 14 days with 7 days recovery (21 day cycle)
  Other Names: TLN-4601

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose (MTD) and the recommended dose for future studies of ECO-4601 administered as a continuous IV infusion for 14 days with 7 days recovery (21 day cycle) in patients with histologically confirmed solid tumors (high grade glioma, colorectal, lung, breast, ovarian, pancreatic and prostate). This study was also designed to determine the clinical pharmacokinetic profile, safety of multiple cycles of administration, and document the antitumor activity of ECO-4601.

ELIGIBILITY:
Inclusion Criteria:

* Informed about the study and consent to participate in the study
* Clinically or radiologically documented advanced solid malignancy for which no standard therapy is available, or which has failed standard therapy
* Patients with the following solid tumors: high grade glioma, colorectal, prostate, pancreatic, lung, ovarian and breast carcinoma
* Age ≥ 18 years of age
* ECOG ≤ 2
* Laboratory hematology and biochemistry protocol test result abnormalities ≤ Grade 1, graded using NCI CTCAE version 3.0
* Patients with no chemotherapy during the 4 weeks preceding patients' first dose of ECO-4601 (day 1, cycle 1)
* No other anticancer treatment during the study
* Patients can be receiving stable or decreasing dose of steroids within 2 weeks prior to patient's signature of the informed consent
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre
* Previous Therapy

  * Hormonal therapy: Patients may have had prior hormonal therapy provided it is discontinued upon ICF signature
  * Radiation: Patients may have had prior radiation therapy. Patients must have recovered from the acute toxic effects of radiotherapy
  * Previous surgery: Previous surgery is permitted provided that at least 2 weeks have elapsed between major surgery (non-biopsy) and ICF signature

Exclusion Criteria:

* Patients with brain metastases
* Unlikely to comply with protocol or difficulty to understand the purpose of the study
* Life expectancy < 12 weeks
* Clinically significant co-morbid disease, e.g. renal failure, ischemic vascular disease, uncontrolled seizure, dementia
* Any patient with a potentially curable malignancy who has not yet received appropriate standard therapies
* Anti seizure drugs known inducers of cytochrome P450
* Documented HIV, active hepatitis B or C infections
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions, which would not permit the patient to be managed according to protocol
* Pregnant or lactating women; both men and women enrolled on study should be using adequate birth control measures throughout the course of the study. Women of childbearing potential must have a negative serum or urine pregnancy test documented within 14 days prior to registration and at study start
* Inability or refusal to practice contraception during therapy of ECO-4601, unless patient is surgically sterile or woman is postmenopausal for at least 2 years
* Patients who have been treated with any investigational drug within 4 weeks of patient's signature of informed consent form, or who are receiving concurrent treatment with other experimental drugs or anti cancer therapy
* Patients in whom a proper central line cannot be established
* Concomitant therapy with therapeutic coumadin; patients can be transferred to low molecular weight heparin
* Patients on low molecular weight heparin for < 2 weeks prior to ICF signature
* Polysorbate 80 being a major constituent of ECO-4601 and known to cause hypotension, patients with uncontrolled hypotension will be excluded
* Known hypersensitivity to farnesylated dibenzodiazepinone or any of the formulation components

Concomitant Therapy Permitted:

* Patients may receive ongoing supportive and palliative care (eg: pain control) as clinically indicated throughout the study.
* Patients can be treated with corticosteroids if medically needed
* Usage of low molecular weight heparin is allowed
* Anti seizure products are permitted provided they are not inducers of cytochrome P450.

Concomitant Therapy Not Permitted:

* Other anticancer treatment
* Other investigational therapy
* Concomitant therapy with coumadin
* Cytochrome enzyme inducing anti epileptics
* G-CSF, GM-CSF and other growth factors may not be used as a substitute for a scheduled dose reduction; however they may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated at the discretion of the investigator. Use of erythropoietin is allowed if treatment has been initiated for ≥ 2 months. Use of growth factors must be documented on case report forms.
* Hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of ECO-4601
Determination of MTD of ECO-4601
Determination of recommended dose for future studies of ECO-4601

SECONDARY OUTCOMES:
Pharmacokinetics of ECO-4601
Safety of multiple cycles of administration of ECO-4601
Documentation of ECO-4601 antitumor activity as per RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kavan, MD, Ph.D., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital; Benoît Samson, MD, Principal Investigator — Hopital Charles Lemoyne; Gerald Batist, MD, Study Chair — Sir Mortimer B. Davis - Jewish General Hospital
Locations (2):
- Canada (2):
  - Hôpital Charles LeMoyne, Greenfield Park, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec